CLINICAL TRIAL: NCT03348592
Title: Gut Microbiome and p-Inulin in CKD TarGut CKD Study
Brief Title: Gut Microbiome and p-Inulin in CKD - TarGut CKD Study
Acronym: TarGut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: George Washington University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jennifer Gassman, Principal Investigator - Data Coordinating Center, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DK099877-T
Record Dates: First submitted 2017-10-31; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Diseases
Keywords: Microbiome, p-inulin
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This is a 28 week study. Participants take no treatment for 8 weeks, followed by 12 weeks on the pre-biotic p-inulin, followed by no treatment for 8 weeks. The treatment arms are no treatment and the pre-biotic p-inulin. Inulin is derived from chicory root fiber.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oligofructose-enriched inulin (p-inulin) (Experimental): Participants are on no treatment for 8 weeks, then the pre-biotic p-inulin for 12 weeks, then no treatment for 8 weeks. Inulin is derived from chicory root fiber. The dose is 16 grams of p-inulin powder per day.
  Interventions: Dietary Supplement: Oligofructose-enriched inulin (p-inulin); Other: No treatment

INTERVENTIONS:
Dietary Supplement: Oligofructose-enriched inulin (p-inulin)
Other: No treatment — Patients do not take a supplement during the first 8 weeks or the last 8 weeks of the study.

SUMMARY:
The purpose of this Phase 1, 3-period crossover with repeated measures feasibility study is to characterize the gut microbiome of individuals with chronic kidney disease, and to explore effects of p-inulin on the gut microbiome. The nature of the study will provide information about the feasibility of stool sample collection for future multicenter studies of the gut microbiome.

DETAILED DESCRIPTION:
The overarching hypothesis motivating this exploratory study of variability is that treatment with oligofructose-enriched inulin (p-inulin) will alter the composition and/or function of the gut microbiome, and thereby reduce the generation of gut-derived uremic toxins, improve gut barrier function and attenuate systemic inflammation in CKD patients. In order to design a future clinical trial the following parameters from CKD subjects are needed:

1. Intra-patient variability in the composition and function of the gut microbiome
2. Inter-patient variability in the composition and function of the gut microbiome
3. Impact of p-inulin on the composition and function of the gut microbiome
4. Tolerability of p-inulin administration
5. Feasibility of collecting stool samples in this patient population

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with eGFR 15.0 to 50.0 ml/min/1.73 m2 as estimated by the CKD-EPI equation
2. Albuminuria greater than 300 mg/g creatinine (by spot urine test) if eGFR is ≥45 ml/min/1.73 m2
3. Age ≥ 18 years
4. For women of childbearing potential, willingness to use a highly effective method of birth control for up to 4 weeks after the last dose to study drug. See Section 4.2.1 for definition of childbearing potential and acceptable methods of birth control
5. Ability to provide informed consent

Exclusion Criteria:

1. Use of pre- or pro-biotics during the past 2 months
2. Consumption of probiotic yogurt during the past 2 weeks
3. Use of antibiotics within the past 3 months if the patient received a single course of antibiotic. If the patient received more than one course of antibiotic treatment, we will wait for 6 months prior to inclusion.
4. Presence of HIV infection, chronic wound infection and osteomyelitis
5. Presence of or treatment for periodontal infection
6. Inflammatory bowel disease, chronic diarrhea, current C. difficile infection
7. Cirrhosis or chronic active hepatitis
8. Treatment with immunosuppressive medications in the past 6 months or more than a week of treatment with prednisone >10 mg in the last 3 months
9. Treatment with proton pump inhibitors within the last one month
10. Anticipated initiation of dialysis or kidney transplant within 9 months
11. Acute on chronic kidney disease
12. Expected survival < 9 months Do not disclose or use except as authorized by the Pilot Clinical Trials in CKD Consortium.
13. Pregnancy, anticipated pregnancy, or breastfeeding
14. Incarceration
15. Participation in another intervention study
16. Severe anemia defined as hemoglobin <9.0 g/dl any time during the last 3 months
17. Patients in whom frequent blood sampling may be difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Microbial composition of stool | Stool is collected weekly for 28 weeks
  Microbial taxonomy will be assigned using Ribosomal Database Project (RDP) for 16S, augmented by analysis of specific sequences using BLAST. The 16S tag sequences will be collected into operational taxonomic units (OTUs) with 97% sequence identity.
Adherence to p inulin prescription | Packets are counted every four weeks during the 12 weeks when the patient is taking p inulin
  Proportion of packets taken vs packets prescribed by packet count

SECONDARY OUTCOMES:
butyrate | Collected weekly for 28 weeks
  captured by untargeted metabolomics, short chain fatty acid in stool blood and urine
propionate | Collected weekly for 28 weeks
  captured by untargeted metabolomics, short chain fatty acid in stool blood and urine
acetate | Collected weekly for 28 weeks
  captured by untargeted metabolomics, short chain fatty acid measured in stool blood and urine
Trimethylamine N oxide | Collected weekly for 28 weeks
  captured by untargeted metabolomics in stool blood and urine
Choline | Collected weekly for 28 weeks
  captured by untargeted metabolomics in stool blood and urine
Betaine | Collected weekly for 28 weeks
  captured by untargeted metabolomics in stool blood and urine
Indoles | collected weekly for 28 weeks
  Indoxyl sulfate Indoxyl glucuronide 5-hydroxyindole Indole-3-prioonic acid Indole-3-acetic acid captured by untargeted metabolomics in stool blood and urine
Phenols | collected weekly for 28 weeks
  p-cresol sulfate p-Cresol glucuronide Phenyl sulfate Phenyl glucuronide α-N-phenylacetyl-L-glutamine Phenylpropionylglycine Hippuric acid 4-hydroxybenzoate Phenylacetylglycine
  * captured by untargeted metabolomics and quantitated by targeted metabolomics in stool blood urine
polyamines | collected weekly for 28 weeks
  captured by untargeted metabolomics in stool blood and urine
metabolites of urea and creatinine metabolism | collected weekly for 28 weeks
  captured by untargeted metabolomics in stool blood and urine
Allantoin | collected weekly for 28 weeks
  captured by untargeted metabolomics in stool blood and urine
Fructose | collected weekly for 28 weeks
  captured by untargeted metabolomics in stool blood and urine
Cytokines | collected weekly for 28 weeks
  IL-1β IL-2 IL-4 IL-6 IL-10 IL-17 IL-22 TNFα measured by standard ELISA in stool
endotoxin | collected weekly for 28 weeks
  measured by standard ELISA in stool
Myeloperoxdase (MPO) | collected weekly for 28 weeks
  measured by standard ELISA in stool
hsCRP | collected weekly for 28 weeks
  measured by standard ELISA in stool
HMGB1 | collected weekly for 28 weeks
  measured by standard ELISA in stool
TNF-R1 | collected weekly for 28 weeks
  measured by standard ELISA in stool
TNF-R2 | collected weekly for 28 weeks
  measured by standard ELISA in stool
Lipopolysaccharide binding protein (LBP) | collected weekly for 28 weeks
  measured by standard ELISA in stool
sCD14 | collected weekly for 28 weeks
  measured by standard ELISA in stool

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Abbott, MD, MPH, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Jennifer J. Gassman, Ph.D., Principal Investigator — The Cleveland Clinic; Linda F. Fried, MD, MPH, Study Chair — VA Pittsburgh Healthcare System
Locations (1):
- The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03348592/Prot_SAP_000.pdf